CLINICAL TRIAL: NCT05431400
Title: Reducing the Risk of Cardiovascular Diseases in Community-dwelling Adults: an Ambispective Cohort Study
Brief Title: Reduction of Risk for Cardiovascular Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-083
Record Dates: First submitted 2022-06-05; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; Prediction model; Community
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — For the prospective part, serum, plasma, urine and fecal samples will be collected for biochemical tests, biomarker examination and DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To establish and evaluate a new prediction model for assessing cardiovascular disease risk in community-dwelling adults.

DETAILED DESCRIPTION:
This is an ambispective, observational cohort study. In the retrospective part, we will enroll residents from Guangzhou or Foshan who participated in the annual health checks provided by the Chinese National Basic Public Health Service project between January 2015 and December 2019. The demographic characteristics, anthropometric measurements, laboratory assays, medical history, living habits, and medications will be collected through personal electronic health records obtained from the regional chronic disease management platform. In the prospective part, residents who participated in the annual health checks provided by the Chinese National Basic Public Health Service project after January 2020 will be enrolled. In addition to the data collected in the retrospective part, blood, urine and fecal samples and lifestyle questionnaires will be collected for further analysis. All participants will be followed-up till December 2025. A new prediction model for assessing cardiovascular disease risk will be established and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Meet at least one of the following conditions: 1. Age ≥ 65 years; 2. Diabetes mellitus; 3. Hypertension;

Exclusion Criteria:

* Refuse to provide informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-dwelling adults in Guangzhou or Foshan who participated in the annual health checks provided by the Chinese National Basic Public Health Service project.
  To participate in the Chinese National Basic Public Health Service project, one must meet at least one of the following conditions: 1. Age ≥ 65 years; 2. Diabetes mellitus; 3. Hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 5 years
  Major adverse cardiovascular events include all-cause mortality, acute myocardial infarction, coronary heart disease, heart failure and stroke.

SECONDARY OUTCOMES:
Atherosclerotic cardiovascular events | 5 years
  Atherosclerotic cardiovascular events include acute myocardial infarction, coronary heart disease, heart failure and fatal and non-fatal stroke.
All-cause mortality | 5 years
  Defined as any death after enrollment.
Cognitive dysfunction | 5 years
  Defined as Montreal Cognitive Assessment (MoCA) Score < 26 points.
Renal functional deterioration | 5 years
  Evaluated through change in estimated glomerular filtration rate.
Renal replacement therapy and/or death due to acute renal failure | 5 years
Incident atrial fibrillation | 5 years
  Atrial fibrillation is diagnosed according to the 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Jiancheng Xiu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (2):
- China (2):
  - The Fourth People's Hospital of Foshan, Foshan, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No